CLINICAL TRIAL: NCT06191016
Title: Effects of Vagal Nerve Stimulation on Pain Frequency and Intensity in Chronic Migraine
Brief Title: Vagal Nerve Stimulation and Pain Frequency, Intensity in Chronic Migraine
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC01746 Rabia Nasir
Record Dates: First submitted 2023-12-19; First posted 2024-01-05 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Migraine
Keywords: chronic migraine; vagal nerve stimulation; pain intensity and frequency
MeSH Terms: conditions — Migraine Disorders; Pain | interventions — Vagus Nerve Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- nVNS Group (Experimental): Experimental group will receive noninvasive vagal nerve stimulation (nVNS) in addition to prescribed medications
  Interventions: Device: Vagal nerve stimulation; Device: Sham vagal nerve stimulation
- Sham Group (Active Comparator): control will receive sham stimulation to vagal nerve along with prescribed medications.
  Interventions: Device: Vagal nerve stimulation; Device: Sham vagal nerve stimulation

INTERVENTIONS:
Device: Vagal nerve stimulation — Experimental group will receive noninvasive vagal nerve stimulation (nVNS) in addition to prescribed medications
Device: Sham vagal nerve stimulation — control will receive sham stimulation to vagal nerve along with prescribed medications

SUMMARY:
This study is being conducted to address the need for effective and well-tolerated interventions in preventing chronic migraine attacks. Chronic migraines significantly impact the quality of life for individuals suffering from them, often leading to substantial discomfort and impairment. By evaluating the feasibility, safety, and acceptance of noninvasive vagus nerve stimulation (nVNS), researchers aim to determine if this approach can offer a viable solution for alleviating the frequency and severity of chronic migraine episodes. If successful, this study could potentially introduce a promising new treatment option that enhances the well-being and daily functioning of those affected by chronic migraines.

DETAILED DESCRIPTION:
Neuromodulation is a growing field in headache management. Technology ranges from invasive deep brain stimulation (DBS) of the posterior hypothalamus, to minimally invasive percutaneous electrode implantation for occipital nerve stimulation, and noninvasive transcranial magnetic stimulation and transcranial direct current stimulation. Neurostimulation can be particularly useful to those who failed triptans or other prophylactic treatments. The European Headache Federation positioned that a neurostimulation device should only be used in medically intractable headache patient who has been evaluated at a tertiary headache center. Vagus nerve stimulation (VNS), which has demonstrated its antinociceptive potential, may also provide a relief of pain associated with headache

ELIGIBILITY:
Inclusion Criteria:

* Chronic migraine (headache for 15 or more days/month for more than three months), Migraine with/without aura

Exclusion Criteria:

* Mental illness, Photophobic individual, Presence of shunt and/or implant at the cranial region

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2023-12-26 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Structured Headache Diary Data for frequency of migraine | Week 4
  Diaries and calendars make possible to record prospectively the characteristics of every attack and this may reduce the recall bias and increase the accuracy of the description.
Numeric Pain Scale (NPS) for intensity of migraine | Week 4
  NPS was implemented in clinical practice due to its rapidity both verbally and in writing. Due to its convenience, it is common for hospitals to measure pain using the 0 to 10 NPS scale
Multidimensional Pain Inventory (MPI) for migraine impact | Week 4
  The MPI was administered pretreatment. It is a 61-item self-administered questionnaire composed of 12 empirically derived scales designed to measure a patients' experiences of pain, their spouses responses to their pain, and their general activity levels

SECONDARY OUTCOMES:
Migraine-Specific Quality of Life Survey (MSQ 2.1) for quality of life | Week 4
  The MSQOL is a measure to assess the effects of migraine over the longer term on patient well-being over a nonspecified time period, and the MQoLQ is designed to measure the short-term impact of migraine over a 24-hour period following the start of therapy for migraine.

CONTACTS AND LOCATIONS:
Overall Officials: Mirza Obaid Baig, MSPT, Principal Investigator — Riphah International University
Locations (1):
- Pakistan Railway General Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vukovic Cvetkovic V, Jensen RH. Neurostimulation for the treatment of chronic migraine and cluster headache. Acta Neurol Scand. 2019 Jan;139(1):4-17. doi: 10.1111/ane.13034. Epub 2018 Oct 29. PMID 30291633
- [Background] Tassorelli C, Grazzi L, de Tommaso M, Pierangeli G, Martelletti P, Rainero I, Dorlas S, Geppetti P, Ambrosini A, Sarchielli P, Liebler E, Barbanti P; PRESTO Study Group. Noninvasive vagus nerve stimulation as acute therapy for migraine: The randomized PRESTO study. Neurology. 2018 Jul 24;91(4):e364-e373. doi: 10.1212/WNL.0000000000005857. Epub 2018 Jun 15. PMID 29907608
- [Background] Lendvai IS, Maier A, Scheele D, Hurlemann R, Kinfe TM. Spotlight on cervical vagus nerve stimulation for the treatment of primary headache disorders: a review. J Pain Res. 2018 Aug 27;11:1613-1625. doi: 10.2147/JPR.S129202. eCollection 2018. PMID 30214271
- [Background] Martelletti P, Barbanti P, Grazzi L, Pierangeli G, Rainero I, Geppetti P, Ambrosini A, Sarchielli P, Tassorelli C, Liebler E, de Tommaso M; PRESTO Study Group. Correction to: Consistent effects of non-invasive vagus nerve stimulation (nVNS) for the acute treatment of migraine: additional findings from the randomized, sham-controlled, double-blind PRESTO trial. J Headache Pain. 2018 Dec 18;19(1):120. doi: 10.1186/s10194-018-0949-9. PMID 30563446